CLINICAL TRIAL: NCT01359358
Title: Epidemiological Study of Methicillin-resistant Staphylococcus Aureus (MRSA) Isolated From Infected Patients During a Hospital Surveillance Period
Brief Title: Study of Methicillin-resistant Staphylococcus Aureus (MRSA) Isolated From Infected Patients in Brazil
Acronym: MRSABrazil
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Sao Paulo (Other)
Responsible Party: Ilana Lopes Baratella da Cunha Camargo, University of Sao Paulo
Other Study IDs: Novartis IFSC-USP
Record Dates: First submitted 2011-05-20; First posted 2011-05-24 (Estimated); Last update posted 2011-05-24 (Estimated); Status verified 2011-05

CONDITIONS: Methicillin Resistant Staphylococcus Aureus
Keywords: MRSA; MLST; PFGE; Resistance; isolated from colonization

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This project has as general objective to determine if there is any Methicillin-resistant Staphylococcus aureus (MRSA) strain disseminating in the hospital of Belo Horizonte. If this is the case, the investigators will determine if this is an international known strain by typing it by PFGE and MLST.

The detection of mecA gene will be performed by PCR. Their susceptibility profile to several drugs will also be accessed and it will be possible to compare the response to those drugs commonly in use to that of Daptomycin, a new drug available in Brazil.

It will be screened for reduced susceptibility to vancomycin by Macromethod Etest (MET) in order to search for VISA or hetero-VISA. Also, due to the discussions at the literature about mutations in genes that are said to be responsible for reduced susceptibility to vancomycin, the investigators will sequence these genes in all PFGE type strain of this study looking for mutations already described to compare to the screening results.

DETAILED DESCRIPTION:
Multidrug resistant and virulent MRSA strains have been disseminating worldwide and few alternatives of treatment for diseases caused by this pathogen are available. In this study, 36 isolates from colonization or different clinical specimens from infected patients of the Hospital Rizoleta Tolentino Neves will be analyzed. These results will provide important data for doctors and nurses, such as whether there is any strain dissemination or not in the hospital what could suggest an outbreak. It will be performed molecular typing by pulsed field gel electrophoresis (PFGE) and multilocus sequence typing (MLST). The investigators will evaluate the efficiency of several antimicrobials and the frequency of h-VISA and VISA among the Brazilian MRSA. Besides, the investigators will verify the presence of mutation in genes that are involved in resistance mechanisms of VISA. According to the strains profile present in the hospital, if this is suggested that there is a dissemination of some strain, the health professionals can start a more rigid infection control measures in order to decrease the number of cases of nosocomial infection, decreasing the time of hospitalization of patients and, consequently the cost for the hospital.

ELIGIBILITY:
Inclusion Criteria:

* MRSA from infection sites
* MRSA from colonization of the patients who already was infected by MRSA during the time of the study

Exclusion Criteria:

* MRSA from colonization of a patient who has not infection caused by MRSA

Min Age: 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: MRSA from infection or from colonization of a patient who was already infected by MRSA during the time of the study
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2011-07

CONTACTS AND LOCATIONS:
Overall Officials: Ilana L B Camargo, PhD, Principal Investigator — University of Sao Paulo
Locations (1):
- Instituto de Física de Sao Carlos - Universidade de Sao Paulo, São Carlos, São Paulo, Brazil